CLINICAL TRIAL: NCT04637997
Title: Influence of Flat-knitted Compression Stockings Class I and II on the Morphology of Venous Malformations - Is There a Therapeutic Effect?
Brief Title: Influence of Flat-knitted Compression Stockings Class I and II on Venous Malformations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Dr. med. Antje Mükke, Senior physician Dr. med. Antje Mükke, University Hospital Erlangen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VM_Compression
Record Dates: First submitted 2020-11-09; First posted 2020-11-20 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Vascular Malformations; Vascular Malformation Peripheral; Venous Malformation; Vascular Diseases
Keywords: Compression therapy; Compression stockings class I; Compression stockings class II; Short-Form 12 (SF-12); Quality of life; Wearing comfort; Magnetic Resonance Imaging; MRI; Perometre
MeSH Terms: conditions — Vascular Malformations; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a single group study with crossover components. Participants receive randomly and double-blinded either class I compression stockings or class II compression stockings. After four weeks, an exchange of compression classes takes place, so that all participants wear both classes of compression stockings within eight weeks.
Who Masked: Participant, Investigator
Masking Description: Double-blind study. Neither investigator nor patient knows the compression class (class I versus class II) of the compression stockings used in the different investigation periods in this patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group 1 (Other): Wearing of compression stockings class I between Investigation day 28 to 56. Wearing of compression stockings class II between Investigation day 56 to 84.
  Interventions: Device: compression stockings class I; Device: compression stockings class II
- Study group 2 (Other): Wearing of compression stockings class II between Investigation day 28 to 56. Wearing of compression stockings class I between Investigation day 56 to 84.
  Interventions: Device: compression stockings class I; Device: compression stockings class II

INTERVENTIONS:
Device: compression stockings class I — Daily wearing of compression stockings class I for four weeks on the affected extremity.
Device: compression stockings class II — Daily wearing of compression stockings class II for four weeks on the affected extremity.

SUMMARY:
Diseases with vascular malformations are rare and often congenital, affecting patients of all ages. Depending on their extent and localization, they can cause discomfort and, especially if activity is restricted, lead to loss or reduced quality of life.

The therapy is usually reserved for a few specialized centers and includes interventional sclerotherapy as well as conservative therapy by compression with appropriate compression stockings. However, there are currently no study-based recommendations for this approach.

The aim of this study is to prove a therapeutic effect of compression therapy using flat-knitted compression stockings on venous malformations of the extremities and to derive from this a therapy recommendation in connection with an improvement in the health status and quality of life.

For this purpose, patients with a confirmed venous malformation of the upper or lower extremity independent of previous therapy will be included. We will investigate patients with epi- and/or subfascial localization of the venous malformation independent of the local extent (cross-articular or not).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed venous malformation of the upper/lower extremity independent of previous therapy with epi- and/or subfascial localization of the venous malformation independent of the local extent (cross-articular or not)
* Compression stocking can be put on independently or by the parents
* Written declaration of consent present

Exclusion Criteria:

* Lack of compliance, patient is not available for control appointments
* Additional drug therapy (anticoagulation) for extensive venous malformations with threatening thromboembolic complications
* Known allergic reaction/intolerance to components of flat-knitted compression stockings
* Pregnancy
* Rejection of the study participation by the patient
* Contraindications for the planned MRI examination (pacemakers, implants not suitable for MRI, claustrophobia)
* Occurrence of an emergency situation
* Severe heart failure as contraindication for compression therapy
* Peripheral arterial disease as contraindication for compression therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Erlangen, Vascular Surgery, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were informed about the possibility of participating in the study during a routine presentation of the vascular surgery consultation Hours during 01.10.2017-01.12.2018.
Period: Overall Study
Arm/Group | Study Group 1 | Study Group 2
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group 1 | Study Group 2 | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.22 (18.91) | 28.11 (15.5) | 27.17 (24.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 9 | 9 | 18
Affected part of body [Count of Participants; unit: Participants]
  arm | 4 | 1 | 5
  lower limb | 3 | 2 | 5
  upper limb | 2 | 4 | 6
  upper and lower limb | 0 | 2 | 2
Previous therapy [Count of Participants; unit: Participants] — Number of participants in whom therapy has already been performed related to the venous malformation.
  Participants | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Volume Difference of Malformation to Baseline (no Compression) While Wearing Compression Stockings Class I and II Determined by MRI
Description: Determination and comparison of volume difference of the malformation after application of compression stockings class I and II compared to baseline (no compression) measured non-invasively by MRI.
Time Frame: one day
Population: Intention-to-treat population (ITT): all randomized participants that received flat-knitted compression stockings class I and class II after the randomization.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Compression Stockings Class I: Wearing of compression stockings class I on the affected extremity.
- Compression Stockings Class II: Wearing of compression stockings class II on the affected extremity.
Arm/Group | Compression Stockings Class I | Compression Stockings Class II
Number analyzed (Participants) | 18 | 18
ml | 16.38 (18.28) | 23.7 (25.67)

2. Primary Outcome: Volume Difference of the Affected Extremity to Baseline (no Compression) While Wearing Compression Stockings Class I and II Determined by Perometre
Description: Determination and comparison of volume difference of the affected extremity after application of compression stockings class I and II compared to baseline (no compression) measured non-invasively by perometre.
Time Frame: one day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Compression Stocking Class I: Daily wearing of compression stockings class I for four weeks on the affected extremity.
Arm/Group | Compression Stocking Class I | Compression Stockings Class II
Number analyzed (Participants) | 18 | 18
ml | 124 (351.09) | 90.22 (226.7)

3. Secondary Outcome: Difference Between Quality of Life at Baseline (no Compression at Day 28) and Compression Classes I and II by Short Form-12 (SF-12) Health Survey at Day 56 or 84
Description: SF-12v2 (SOEP-Version 2004) scale is a generic, multipurpose short-form survey with 12 questions selected from the SF-36 Health Survey which, when combined, scored and weighted, results in two scales of mental (MCS) and physical (PCS) functioning and overall health-related quality of life.
  A higher value indicates a better quality of life of the patient. The scores range from 0 to 100. The overall mean for each scale is 50 points and the standard deviation is 10 points in the SOEP sample.
Time Frame: up to two months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Compression Stockings Class I: Difference between Quality of life after daily wearing of compression stockings class I for four weeks on the affected extremity.
- Compression Stockings Class II: Difference between Quality of life after daily wearing of compression stockings class II for four weeks on the affected extremity.
Arm/Group | Compression Stockings Class I | Compression Stockings Class II
Number analyzed (Participants) | 18 | 18
units on a scale
  PCS | 1.9505 (7.2323) | 3.3461 (7.321)
  MCS | 1.0922 (9.6244) | 0.1778 (6.865)
  Overall Health-related Quality of life | 1.5214 (4.24) | 1.762 (3.164)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 18 months during the enrollment, inclusion and investigation period of participants.
Description: During the whole Investigation period there were no participants at Risk for All-Cause Mortality because no potentially life-threatening diagnosis, treatment or therapy was performed. Especially there was no use of drugs, contrast agent or other potentially allergy triggering procedures. All procedures related to the study have been performed non-invasively. Nevertheless, all-cause mortality was monitored.
Groups:
- Compression Stockings Class I: Wearing of compression stockings class I on the effected extremity for four weeks between Investigation day 28 to 56 or between Investigation day 56 to 84.
- Compression Stockings Class II: Wearing of compression stockings class II on the effected extremity for four weeks between Investigation day 28 to 56 or between Investigation day 56 to 84.
Arm/Group | Compression Stockings Class I | Compression Stockings Class II
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT04637997/Prot_SAP_000.pdf